CLINICAL TRIAL: NCT04858854
Title: Effect of Broccoli Sprout Extract in Patients With Chronic Kidney Disease With Diabetes Type 2
Acronym: INITIATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Lantmännen (Unknown)
Responsible Party: Principal Investigator, Peter Stenvinkel, Principal investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-06468
Record Dates: First submitted 2021-04-09; First posted 2021-04-26 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Chronic Kidney Disease Stage 3B; Chronic Kidney Disease stage4; Diabetes Mellitus, Type 2
Keywords: Sulforaphane; Nutrition; Glucose control
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — sulforaphane

STUDY DESIGN:
Intervention Model Description: This is a multicentre randomized double-blinded controlled trial lasting 20 weeks with two study periods. The first 12 weeks will constitute a treatment period with BSE (BSE group) or placebo (Control group) depending on the randomization of the group allocation. After that, patients from both groups will be followed for another eigth weeks, called post-study observational period.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BSE group (Broccoli sprout group) (Active Comparator): The BSE Group will receive 50 µmmol/day of sulforaphane administered by BSE (Lantmännen®) from week 0 to week 4. If no side-effects are reported, the sulforaphane dose will increase to 100 µmmol/day from week 5 to week 8 and in the absence of side-effects, the dose will increase to 150 µmmol/day from week 9 to week 12.
  Interventions: Other: Sulforaphane, administered as Broccoli sprout extract
- Control group (Placebo Comparator): The Control Group will receive a placebo (maltodextrin sprayed with copper-chlorophyllin) for 12 weeks.
  Interventions: Other: Sulforaphane, administered as Broccoli sprout extract

INTERVENTIONS:
Other: Sulforaphane, administered as Broccoli sprout extract — Patients will randomized to BSE or Control Group. The group BSE will receive the sulforaphane, administered as broccoli sprout extract for 12 weeks. The dose will increase every four weeks if no side-effects are reported (50 µmmol/day; 100 µmmol/day and 150 µmmol/day, respectivelly). The Control group will receive a placebo (maltodextrin sprayed with copper-chlorophyllin) for the same period (12 weeks). The BSE/placebo will be administered as powder provided in 10 ml of water in the morning in a double-blind manner as dry mixtures in sealed portion size bags of similar shape and size.

SUMMARY:
This research project aims to test if sulforaphane, administered as broccoli sprout extract (BSE) can ameliorate glucose control in adult patients with chronic kidney disease (CKD) and DM 2 with GFR > 15 < 45 ml/min/1.73 m2. The glucose control will be evaluated by the oral glucose tolerance test. Moreover, as a secondary aim, we will investigate the role of sulforaphane in improving other signs of metabolic derangements present in this group of patients, including oxidate stress, proteinuria, inflammation and a decrease in the production of uremic toxins from the gut microbiota. This a multicentre randomized double-blinded controlled trial including 100 adult patients with CKD and glomerular filtration rate (GFR) between 15 and 29 ml/min/1.73m2, DM type 2, age > 18 years old. Patients will be randomized into BSE group or Placebo group. Both groups will be followed for 20 weeks: The first 12 weeks patients will receive the BSE or Placebo and, the next 8 weeks, both groups will be followed with no intervention to observe the changes in the primary and secondary outcomes. Patients randomized to BSE Group will receive 50 µmmol/day of sulforaphane administered as BSE (Lantmännen®) from week 0 to week 4. If no side-effects are reported, the sulforaphane dose will increase to 100 µmmol/day from week 5 to week 8 and in the absence of side-effects, the dose will increase to 150 µmmol/day from week 9 to week 12. Blood and urine samples and OGTT (in non-insulin dependent patients) will be performed at week 0, 12 and 20. On week 4 and 8 blood drawn for partial exam will be performed. The BSE and the placebo (maltodextrin sprayed with copper-chlorophyllin) will be administered as powder provided in a double-blind manner as dry mixtures in sealed portion size bags of similar shape and size. Randomization will be done using a computer-based block randomization algorithm. Comparisons between the primary and secondary studied variables will be done with two-way analysis of variance (ANOVA) with repeated measures for normally distributed variables. Variables that can interfere with the glycemic control, such as changes in the dosage of hypoglicemiants agents and insulin during the intervention will be controlled in the analysis. Those non-normally distributed will be log transformed aiming to normalize the distribution. All test will consider a P<0.05 for statistical significance. The software Stata will be used for the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a GFR 15-45 ml/min/1.73 m2, DM type 2, age >18 years old, able to read and understand Swedish.

Exclusion Criteria:

* Use of metformin, use of warfarin, levels of ASAT, ALAT more than three times the upper limit at screening or at any subsequent visit, kidney transplantation, inflammatory bowel disease, celiac disease, malignant diseases (except skin basalioma) in the previous 3 years, and any other condition that the treating doctor believes is contraindicated; allergy to broccoli; participation in another clinical trial which may affect the outcome of the present study; not to understand the study information.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
Fasting serum glucose | Baseline, Week 12
  Change in fasting serum glucose from baseline at week 12

SECONDARY OUTCOMES:
C-reactive protein (CRP) | Baseline, Week 12 and Week 20
  Inflammatory marker
Interleukin-6 (IL6) | Baseline, Week 12 and Week 20
  Inflammatory marker
Tumor necrosis alpha (TNF) | Baseline, Week 12 and Week 20
  Inflammatory marker
Interleukin 10 | Baseline, Week 12 and Week 20
  Inflammatory marker
Advanced oxidation protein products (AOPP) | Baseline, Week 12 and Week 20
  Oxidative stress
8-hydroxydeoxyguanosine (8-OHdG) | Baseline, Week 12 and Week 20
  Oxidative stress
Urinary albumin creatinine ratio (ACR) | Baseline, Week 12 and Week 20
  Proteinuria
Indoxyl-sulfate (IS) | Baseline, Week 12 and Week 20
  Uremic toxins
Trimethylamine N-oxide (TMAO) | Baseline, Week 12 and Week 20
  Uremic toxins
P-cresyl sulfate (IPC) | Baseline, Week 12 and Week 20
  Uremic toxins
Oral glucose tolerance test | Baseline, Week 12 and Week 20
  Performed in patients not using insulin at the local participating Hospital Chemical
Fasting HbA1c | Baseline, Week 12, Week 20 and week 20
  Fasting HbA1c
Fasting insulin | Baseline, Week 4, Week 8, Week 12 and Week 20
  Fasting insulin

CONTACTS AND LOCATIONS:
Overall Officials: Peter x Stenvinkel, MD, Principal Investigator — Karolinska Institutet; Carla Avesani, PhD, Study Chair — Karolinska Institutet; Marie Evans, MD, Study Director — Karolinska Institutet
Locations (12):
- Sweden (12):
  - Gävle Hospital, Gävle
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Linköpings universitet, Linköping
  - Skånes University Hospital Sus, Lund
  - Skånes universitetssjukhus, Malmo
  - Karolinska Institutet, Stockholm
  - Danderyds sjukhus AB, Stockholm
  - Norrlands Universitetssjukhus, Umeå
  - Akademiska sjukhuset, Uppsala
  - Hallands Hospital Varberg, Varberg
  - Västmanlands Hospital Västerås, Västerås
  - Västervikssjukhus, Västervik

IPD SHARING:
Plan to Share IPD: No